CLINICAL TRIAL: NCT03623932
Title: Contribution of a Non Medicamentous Approach by Hypnosis on Quality of Life in Crohn Disease
Acronym: HYPNOCROHN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 38RC17.298
Record Dates: First submitted 2018-07-04; First posted 2018-08-09 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Tumor Necrosis Factor-alpha; Hypnosis

STUDY DESIGN:
Intervention Model Description: Prospective study, monocentric, controlled, randomized, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immunosuppressor/TNFalpha (Active Comparator): Standard treatment with immunosuppressor and/or anti-TNFalpha treatment.
  Interventions: Drug: immunosuppressor/TNFalpha
- Hypnosis + Standard Treatment (Experimental): Standard treatment with immunosuppressor and/or anti-TNFalpha treatment in addition to hypnosis parallel treatment.
  Interventions: Behavioral: Hypnosis

INTERVENTIONS:
Drug: immunosuppressor/TNFalpha — Standard Treatment : immunosuppressor/TNFalpha as in standard practice
  Arms: immunosuppressor/TNFalpha
Behavioral: Hypnosis — 8 hypnosis group sessions during 2 months
  Arms: Hypnosis + Standard Treatment

SUMMARY:
Evaluation of hypnosis therapy efficacy in addition to pharmacologic standard treatment of Croh disease during remission by the evaluation of quality of life;

DETAILED DESCRIPTION:
Crohn disease is defined as an inflammatory chronic disease of the bowel characterize by intermittent flare-ups and remission periods.

Crohn disease is due to genetic and environmental factors such as stress. Stress is an important aggravation factor of the disease symptoms which can stop a remission period and induce a relapse into a flare-up period.

Hypnosis is a non-medicinal technic which already show efficacy in the treatment of functional digestive troubles. These diseases are bio/psycho/social models such as Crohn disease.

Hypnosis can reduce visceral pain sensibility, reduce stress and reduce pro-inflammatory cytokines liberation into intestinal mucosa.

Though, only few data are available on hypnosis interest in the treatment of Crohn disease and inflammatory bowel diseases as it is often isolated clinical case report.

One study on patients with rectocolitis in remission period has been done recently and show that hypnosis increased the duration of the remission period.

The principal objective of this study is to evaluate hypnosis efficacy in term of quality of life for patients with Crohn disease during remission.

ELIGIBILITY:
Inclusion Criteria:

* patient with ileal or colic Crohn disease
* stable treatment for Crohn disease
* clinical and biologic remission (normal C reactive protein and fecal calprotectin < 100 µg/g)
* patient living in Grenoble area
* informed consent form
* social security affiliation

Exclusion Criteria:

* Person under legal protection (articles L1121-5 and L1121-8 of Public health code)
* Person in exclusion period of another study
* Hypnosis contraindication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-13 (Actual); Primary Completion 2021-11-12 (Estimated); Study Completion 2021-11-13 (Estimated)

PRIMARY OUTCOMES:
Mid term hypnosis efficacy with IBDQ | 6 months
  Efficacy evaluation of hypnosis 6 months after the beginning of hypnosis sessions on the quality of life with Inflammatory Bowel Disease Questionnaire (IBDQ)

SECONDARY OUTCOMES:
Short term hypnosis efficacy with IBDQ | 3 months
  Efficacy evaluation of hypnosis 3 months after the beginning of hypnosis sessions on the quality of life with Inflammatory Bowel Disease Questionnaire (IBDQ)
Disease acceptance with ICQ-18 | 3 months and 6 months
  Impact of hypnosis on the disease acceptance short and mid term with the Evolution of the Illness Cognition Questionnaire for chronic disease
Clinical score with Harvey-Bradshaw Index short and mid term | 3 months and 6 months
  Evolution of the clinical score short and mid term with Harvey-Bradshaw Index
Vagal tonus with electrocardiogram | 3 months and 6 months
  Evolution of the vagal tonus with electrocardiogram short and mid term
Inflammatory status with C Reactive Protein | 3 months and 6 months
  Evolution of the C Reactive Protein concentration in the plasma
Stress with Perceived Stress Scale | 3 months and 6 months
  Evolution of stress status short and mid term with Perceived Stress Scale which goes from 10 to 50. Lower values represent better outcome.
Fatigue with Multidimensional Fatigue Inventory | 3 months and 6 months
  Evolution of fatigue status short and mid term
Long term hypnosis efficacy | 12 months
  Efficacy evaluation of hypnosis 12 months after the beginning of hypnosis sessions on the quality of life with Inflammatory Bowel Disease Questionnaire (IBDQ) which goes from 32 to 224. Higher values represent better outcome.
Clinical score with Harvey-Bradshaw Index long term | 12 months
  Evolution of the clinical score long term with Harvey-Bradshaw Index

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Grenoble, France

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391